CLINICAL TRIAL: NCT03435900
Title: Intraperitoneal Administration of Fosfomycin, Metronidazole and Molgramostim Versus Intravenous Conventional Antibiotics for Perforated Appendicitis - a Pivotal Quasi-randomized Controlled Trial
Brief Title: Intraperitoneal Administration of Fosfomycin, Metronidazole and Molgramostim Versus Intravenous Antibiotics for Perforated Appendicitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Siv Fonnes, MD, PhD-student, Herlev Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEH-SF-02
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Appendicitis Perforated
MeSH Terms: conditions — Appendicitis | interventions — Metronidazole; regramostim

STUDY DESIGN:
Intervention Model Description: Quasi-randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Drug: Combination of fosfomycin, metronidazole and rhGM-CSF (administered together intraperitoneally) and three days of antibiotics p.o.
- Control group (Active Comparator)
  Interventions: Drug: Standard antibiotics intravenously

INTERVENTIONS:
Drug: Combination of fosfomycin, metronidazole and rhGM-CSF (administered together intraperitoneally) and three days of antibiotics p.o. — All drugs will be administered together intraperitoneally at the end of the surgery after the appendix has been removed. Hereafter, the intervention group will receive three days of orally administered antibiotics: 500 mg amoxicillin combined with 125 mg clavulanic acid and 500 mg metronidazole. These doses will be administered three times daily.
  Arms: Intervention group
Drug: Standard antibiotics intravenously — 4 g piperacillin/500 mg tazobactam and 1 g metronidazole administered intravenously during surgery followed by 4 g piperacillin/500 mg tazobactam and 500 mg metronidazole administered intravenously three times daily for three days.
  Arms: Control group

SUMMARY:
The objective of this trial is to evaluate if intraoperative intraperitoneal administration of fosfomycin, metronidazole and recombinant human granulocyte-macrophage colony-stimulating factor (rhGM-CSF) followed by oral antibiotic for three days is as effective as the current intravenous antibiotic treatment given during and three days after appendectomy for perforated appendicitis. The primary outcome is the total length of hospital stay, defined as the number of hours in hospital after end of operation and until 30-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Suspicion of acute appendicitis and planned for diagnostic laparoscopy and eventual laparoscopic appendectomy
* Perforated appendicitis (diagnosed during surgery by the surgeon)
* Negative p-HCG (women)
* Written informed consent after written and verbal information (preoperatively for the intervention group and postoperatively for the control group)

Exclusion Criteria:

* Cannot understand, read or speak Danish
* Previous allergic reaction to fosfomycin, metronidazole, rhGM-CSF, or penicillins e.g. piperacillin or amoxicillin
* Diagnostic laparoscopy revealing normal appendix not requiring an appendectomy or appendicitis without perforation
* Other intra-abdominal pathology requiring surgical intervention at the same operation
* Known renal or hepatic disease or biochemical evidence at the time of admission
* Known hematologic disease in current medical treatment
* American Society of Anesthesiologists (ASA) physical status ≥4 (a patient with severe systemic disease that is a constant threat to life)
* Body weight >110 kg
* Surgery converted to open appendectomy
* Anticipated compliance problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Total length of hospital stay | From end of surgery until 30-days follow-up
  in hours

SECONDARY OUTCOMES:
Gastrointestinal Quality of Life Index (GIQLI) | 10 days (±2 days) and 30 days (±3 days) postoperatively
  A disease-specific questionnaire validated in Danish is collected at 10 days postoperatively (±2 days) and at 30 days postoperatively (±3 days)
Side effects | Within 24 hours after surgery and 10 days (±2 days) postoperatively
  Number and description. A questionnaire regarding side effects is collected within the first 24 hours after surgery and at 10 days postoperatively (±2 days)
Postoperative complications | From end of surgery until 30-days follow-up
  Number. According to the Clavien-Dindo grading
Surgical site infections requiring surgical drainage | From end of surgery until 30-days follow-up
  It is defined as deep incisional surgical site infection according to Centre for Disease Control and Prevention (CDC)
Intraabdominal abscesses requiring drainage | From end of surgery until 30-days follow-up
  Number. It is defined as an organ/space surgical site infection according to CDC
Readmissions | From end of surgery until 30-days follow-up
  Number. Only readmissions related to the surgery will be registered; e.g. admission and treatment of a non-related condition will not be registered.
Reoperations | From end of surgery until 30-days follow-up
  Number. Only reoperations related to the appendectomy will be registered.
Time to return to normal activities | From end of surgery until 30-days follow-up
  Time period in days. The date is defined at the time point at which the participant could return to normal daily activities.
Period of sick leave "absence from work" | From end of surgery until 30-days follow-up
  Time periode in days. The parameter is defined as the number of days from the operation to the time point at where the participant returned to work or school.
Costs | From end of surgery until 30-days follow-up
  The estimated total costs of admission, surgery, possible complications, reoperations etc. in the two treatment groups.
Adverse events | From end of surgery until 30-days follow-up
Microbiological flora and susceptibility | From end of surgery until 30-days follow-up
  Number and type of positive specimens. If participants have a postoperative infectious complication.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Department of Surgery, Bispebjerg Hospital, Copenhagen
  - Department of Surgery, Herlev Hospital, Herlev

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fonnes S, Roepstorff S, Holzknecht BJ, Olesen CS, Olsen JHH, Schmidt L, Alder R, Gamborg S, Rasmussen T, Arpi M, Jorgensen LN, Rosenberg J. Shorter Total Length of Stay After Intraperitoneal Fosfomycin, Metronidazole, and Molgramostim for Complicated Appendicitis: A Pivotal Quasi-Randomized Controlled Trial. Front Surg. 2020 May 5;7:25. doi: 10.3389/fsurg.2020.00025. eCollection 2020. PMID 32432123